CLINICAL TRIAL: NCT03312647
Title: Adverse Drug Reactions to Antituberculosis Drugs in the Treatment of Latent Tuberculosis Infection in Korean Health Care Workers
Brief Title: Adverse Drug Reactions to Anti-TB Drugs in the Treatment of Latent Tuberculosis Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Dong Won Park, Assistant professor, Hanyang University
Other Study IDs: HYUMC_CM_002
Record Dates: First submitted 2017-06-18; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Latent Tuberculosis Infection
Keywords: Adverse Drug Reaction; Latent Tuberculosis Infection; Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis; Drug-Related Side Effects and Adverse Reactions; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Latent tuberculosis infection: Identified subjects with latent tuberculosis infection (LTBI) using whole-blood interferon-r release assays. All enrolled subjects were treated with one of the recommended regimens for LTBI treatment: 9 months of isoniazid, 4 months of rifampin and 3 months of isoniazid plus rifampin. Blood, urine sampling, and monitoring frequencies of adverse reactions of anti-TB drugs were performed.

SUMMARY:
The investigators aim to study the prevalence of adverse reactions of anti-tuberculosis (TB) drugs in latent tuberculosis infection (LTBI), and determine the risk factors of anti-TB drug-related toxicity in LTBI in Korean health care workers(HCWs).

DETAILED DESCRIPTION:
Further study details as provided by Hanyang University Hospital

This study is prospective study of newly diagnosed LTBI in HCWs at Hanyang University Hospital, a tertiary referral hospital in South Korea, between 2017 and 2018. This study aimed to identify the prevalence of adverse reactions of treatment regimen for LTBI. The diagnosis of LTBI was made on the basis of interferon-gamma releasing assay. Information on demographic characteristics, comorbidity and treatment outcomes was collated from questionnaires. Treatment regimen for LTBI was chosen by patients' preference among 3 months of INH(isoniazid) plus RFP(rifampin), 4 months of RFP and 9 months of INH. All PTB patients were observed 2 weeks after the initiation of medication, and monthly thereafter, and were asked about any drug side effects at these visits. Serious adverse drug reaction (ADR) was defined as any severe side effect that resulted in discontinuation or change (either temporally or permanently) of anti-TB medication, and/or directly resulted in hospitalization. Drug-induced hepatitis was defined as liver transaminases more than three times higher than the upper limit of normal in the presence of symptoms such as anorexia, nausea, vomiting, or abdominal pain, or transaminases more than five times the upper limit of normal without symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or more
* Identified latent tuberculosis infection (LTBI) in Korean health care workers, using whole-blood interferon-r release assays

Exclusion Criteria:

* Subjects who do not want to participate the present study
* Subjects who do not receive LTBI treatment due to abnormal liver function test (i.e, liver cirrhosis etc)
* Subjects with history of previously treated TB
* Subjects with active tuberculosis infection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with latent tuberculosis infection (LTBI) using whole-blood interferon-r release assays in Korean health care workers.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The numbers of adverse drug reactions (ADR) during LTBI treatment | one year
  All events of adverse drug reactions (ADR) were reported using the clinical signs, symptoms, and liver chemistry at predefined intervals (two weeks after the initiation of anti-TB drugs, and monthly thereafter).

SECONDARY OUTCOMES:
The numbers of severe ADR during LTBI treatment | one year
  Among all ADR, serious ADR was defined as any severe side effect that resulted in discontinuation or change (either temporally or permanently) of anti-TB drugs, and/or directly resulted in hospitalization. Drug-induced hepatitis was defined as liver transaminases more than three times higher than the upper limit of normal (γ-glutamyl transpeptidase (γ-GT) >69 U/L; serum glutamic oxaloacetic transminase (SGOT) >54 U/L; serum glutamic pyruvic transminase (SGPT) >60 U/L) in the presence of symptoms such as anorexia, nausea, vomiting, or abdominal pain, or transaminases more than five times the upper limit of normal without symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Heon Kim, MD, PhD., Study Director — Department of Internal Medicine, Hanyang University College of Medicine, Seoul, Korea
Locations (1):
- Sang-Heon Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No